CLINICAL TRIAL: NCT05327543
Title: Effects of Two Different Online Yoga Interventions on the Quality of Life of Breast Cancer Patients Compared With Waiting List - a Three-arm Randomized Controlled Trial
Brief Title: Effects of Online Yoga on the Quality of Life of Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. Andreas Michalsen, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YOMA
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Breast Neoplasms; Cancer
Keywords: Yoga
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Iyengar yoga (Experimental): Intervention group 1 receives an Iyengar yoga intervention online in a group setting, based on the internationally renowned yoga school of B.K.S. Iyengar, which in the context of this study primarily includes physical and relaxation exercises.
  Interventions: Behavioral: Iyengar Yoga
- Meditative yoga (Experimental): Intervention group 2 receives an Integrative yoga intervention online including physical and meditation exercises as well as ideologically neutral explanations of the ethical aspects of Yoga.
  Interventions: Behavioral: Meditative Yoga
- Waitlist Control Group (No Intervention): Group 3 consists of a waitlist control group. Participants will be offered the opportunity to attend a yoga intervention after 4 months. The patients in this waiting list control group are allowed to choose the yoga course after 4 months.

INTERVENTIONS:
Behavioral: Iyengar Yoga — Iyengar Yoga focuses on the correct alignment of the body while practicing the physical exercises of yoga. Props are used to support the body in finding the right alignment. Relaxation is also part of this intervention. Participiants receive 1x90 min guided yoga class per week for 8 weeks and are encouraged to continue their practice at home daily for at least 30 minutes.
  Arms: Iyengar yoga
Behavioral: Meditative Yoga — Meditative Yoga in the context of this study means practicing the physical exercises of yoga as well as meditation. Additionally, each week one of the yamas/niyamas, which are ethical principles to live by in the Yoga philosophy, will be presented at the beginning of each class and will form the theme of the class. Participants receive 1x90 min guided yoga class per week for 8 weeks and are encouraged to continue their practice at home daily for at least 30 minutes.
  Arms: Meditative yoga

SUMMARY:
This study investigates the effects of two different online yoga interventions on the health-related quality of life in breast cancer patients. Qualitative and quantitative data will be collected.

DETAILED DESCRIPTION:
In this randomized controlled trial breast cancer patients will be randomized into three treatment arms:

* Intervention group 1 will receive an Iyengar yoga intervention online in a group setting, based on the internationally renowned yoga school of B.K.S. Iyengar, which in the context of this study mainly includes physical and relaxation exercises.
* Intervention group 2 will receive a meditative yoga intervention online including physical and meditation exercises and also ideologically neutral explanations of the ethical aspects of yoga.
* Group 3 consists of a waiting list control group, combined with the offer to participate in a yoga intervention after 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-metastatic breast cancer (TNM stage I-III) up to 5 years after diagnosis
* Primary therapy completed for at least 3 months
* Limitation of the quality of life due to the cancer (indication of at least 4 out of 10 points on the numerical analogue scale)
* Willingness to participate in the study and signed informed consent.

Exclusion Criteria:

* Current or planned chemotherapy, radiation or surgery
* Severe physical or psychopharmacologically treated psychiatric comorbidity due to which a patient is unable to participate in the study
* Pregnancy/breastfeeding
* Participation in other clinical trials with behavioral, psychological, or complementary medicine interventions
* Immobility or limitation for gymnastic exercise due to orthopedic, neurologic, or other medical cause
* regular meditation practice >2x/month
* regular yoga practice >2x/month

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) | Date of inclusion (baseline), after 8 weeks
  Assessing full scale, range 0-40, higher score meaning a better outcome

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) | Date of inclusion (baseline), after 8 weeks, after 16 weeks, after 24 weeks
  Assessing full scale, range 0-40, higher score meaning a better outcome
Functional Assessment of Cancer Therapy: Fatigue (FACIT-F) | Date of inclusion (baseline), after 8 weeks, after 16 weeks, after 24 weeks
  Assessing full scale, range 0-52, higher score meaning a better outcom
Perceived Stress Scale (PSS-10) | Date of inclusion (baseline), after 8 weeks, after 16 weeks, after 24 weeks
  Assessing full scale, range 0-40, lower score meaning a better outcome
Flourishing Scale (FS-D) | Date of inclusion (baseline), after 8 weeks, after 16 weeks, after 24 weeks
  Assessing full scale, range 8-56, higher score meaning a better outcome
Self-Compassion Scale (SCS-D) | Date of inclusion (baseline), after 8 weeks, after 16 weeks, after 24 weeks
  Mean score of 12 items, range 1-5, higher score meaning a better outcome
Self-Efficacy Scale (ASKU) | Date of inclusion (baseline), after 8 weeks, after 16 weeks, after 24 weeks
  Mean score of 3 items, range 1-5, higher score meaning a better outcome
Sociodemographic measures | Date of inclusion (baseline)
  Age, education level, personal income, household income, employment status, job description, marital status, household members, days of sick leave past 3 months
Behavioral questions: cigarettes | Date of inclusion (baseline), after 8 weeks, after 16 weeks, after 24 weeks
  Number of cigarettes on average per day in the last month
Behavioral questions: alcohol | Date of inclusion (baseline), after 8 weeks, after 16 weeks, after 24 weeks
  Number of alcoholic beverages on average per week in the last month
Expectation question | Date of inclusion (baseline)
  expectation of effectiveness of the intervention on a 5-point likert scale, how they expect to handle the intervention on a 5-point likert scale, higher score meaning better outcome
Behavioural question | Date of inclusion (baseline), after 8 weeks, after 16 weeks, after 24 weeks
  diet
Behavioural question 2 | Date of inclusion (baseline)
  Practice of other mindfulness practices besides Yoga
Behavioural question 3 | Date of inclusion (baseline)
  Yoga styles were practiced before
Behavioural question 4 | Date of inclusion (baseline)
  If and how often yoga is practiced regularly
Functional Assessment of Cancer Therapy - General (FACT-G) | Date of inclusion (baseline), after 8 weeks, after 16 weeks, after 24 weeks
  Assessing full scale, range 0-108, higher score meaning a better outcome
Yama/Niyama Questionnaire - YaNiQ | Date of inclusion (baseline), after 8 weeks, after 16 weeks, after 24 weeks
  Assessing full scale, range 0-100, higher score meaning a better outcome
Hospital Anxiety and Depression Scale (HADS) | Date of inclusion (baseline), after 8 weeks, after 16 weeks, after 24 weeks
  Assessing full scale, range 0-42, lower score meaning a better outcome

OTHER OUTCOMES:
Qualitative interviews | 8 weeks after inclusion
  Qualitative assessment will be carried out in qualitative interviews in 20 patients participating in the study. The interviews will be recorded, transcribed and analyzed with qualitative content analysis.
Heart Rate Variability (HRV) | Date of inclusion (baseline), after 8 weeks
  24h measuring by Faros 180

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, State of Berlin, Germany